CLINICAL TRIAL: NCT03521310
Title: Immediate Parent -Infant Skin-to-Skin Study (IPISTOSS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Continued randomization was questioned on ethical grounds after the WHO iKMC study reported mortality reduction in May 2021. The DSMB recommended to stop the trial after reviewing a preliminary data analysis because of benefit of the intervention.
Sponsor: Björn Westrup, MD PhD (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor-Investigator, Björn Westrup, MD PhD, Co-director of Karolinska NIDCAP Training and Research Center, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPISTOSS
Record Dates: First submitted 2018-02-20; First posted 2018-05-11 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Prematurity
Keywords: IPISTOSS; Skin to skin; SSC; Neonatal; kangaroo mother care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin-to-skin Contact group (Experimental): Neonates in gestational age between 28+0 - 32+6 will get continuous Skin-to-skin contact with one parent/caregiver the first 6 hours after birth and as much as possible the first 72 hours after birth.
  Interventions: Procedure: Skin-to-skin
- Conventional care group (Active Comparator): Neonates in gestational age between 28+0 - 32+6 will get Conventional care - incubators, warmers etc - the first 72 hours after birth.
  Interventions: Procedure: Conventional care

INTERVENTIONS:
Procedure: Skin-to-skin — Neonates will get Skin-to-skin Contact with parent/caregiver continuously the first 6 hours after birth and as much as possible the first 72 hours after birth.
  Arms: Skin-to-skin Contact group
Procedure: Conventional care — Neonates will get Conventional care the first 72 hours after birth
  Arms: Conventional care group

SUMMARY:
The World Health Organization recommend all stable low birth weight neonates to have Skin-to-skin-Contact (SSC) after birth. Intermittent SSC is used in Sweden in neonatal units. Observations indicate that SSC makes neonates feel good. However, there is limited research done on SSC treatment on neonates born prior to week 33.

The aim of this study is to investigate whether Skin-to-skin-Contact (SSC) leads to an improved physiological stabilization, altered epigenetic profile and improved longterm psychomotor outcome in neonates born in gestation age between week 28+0 - 32+6. This is a parallel, two-arm, multicentre, randomized controlled superiority trial. The two arms to be compared are a) immediate SSC with one parent/caregiver continous during the first 6 hours after birth and as much as possible during the first 72 hours, and b) conventional method of care during the same time.

ELIGIBILITY:
Inclusion Criteria:

* Born in gestation week plus days 28+0 - 32+6.
* Born at maternity ward at study center
* Consent from parents/caregivers
* Parent or caregiver or substitute are available to start skin-to-skin Contact during the first hour of life.

Exclusion Criteria:

* Born outside the hospital
* Triplets or more
* Known malformation which will require immediate surgical action
* On-going resuscitation or intensive Medical care (mechanic ventilation or inotropy) after the first lifespan

  * Known congenital infection
* Parent/care giver can not communicate in Swedish/Norwegian or English
* Not suited for the study for other reasons (according to the principal investigator)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory stability | After six hours
  Using the Stability of the CardioRespiratory system In the Preterm-score (SCRIP-score). A higher SCRIP score indicates greater physiological stability

SECONDARY OUTCOMES:
Need for respiratory support | After 3 months
  Days in respirator from birth to discharge from hospital
Need for surfactant | After 3 months
  Number of doses of surfactants from birth to discharge from hospital,
Need of Continuous positive airway pressure | After 3 months
  Days in use of Continuous positive airway pressure (CPAP)- from birth to discharge from hospital
Need for oxygen | After 3 months
  Days in use of oxygen from birth to discharge from hospital
Heart Rate Variability | Up to 3-4 months
Body temperature | At 0 hour (postpartum), 1, 2, 3, 4, 5 and 6 hours
  Axillary body temperature
Sepsis episodes | After 3 months
  Number of Sepsis episodes from birth to discharge from hospital, based on the Medical records
Number of Antibiotic treatment | After 3 months
  Number of Days with antibiotic treatment from birth to discharge from hospital based on Medical records
Status of Breast-feeding | Up to12 months
  Status of Breast-feeding according to a specific questionnaire: Index of Breastfeeding (IBS)
Status of Breast-feeding | Up to12 months
  Status of Breast-feeding according to a specific questionnaire: Breastfeeding Self efficacy Questionnaire (BSES)
Status of Breast-feeding | Up to12 months
  Status of Breast-feeding according to a specific questionnaire: Infant Breastfeeding Assessment Tool (IBFAT).
Time to Full enteral nutrition | After 3 months
  Days from birth until Full enteral nutrition
Time in use of Nasogastric tube feeding | After 3 months
  Days from birth in use of Nasogastric tube feeding
Time to recovered birth weight | After 3 months
  Days from birth until recovered birth weight
Weight gain | Up to 12 months
  Weight gain from birth
Epigenetic profiling in buccal cells | Up to 24 months
  Whole-genome methylation analysis and locus specific analysis of selected stress related genes, will be conducted to investigate early, intermediate and long-term epigenetic changes due to the intervention.
Telomere profiling in buccal cells | Up to 24 months
  Whole-genome methylation analysis and locus specific analysis of selected stress related genes, will be conducted to investigate telomere length.
Epigenetic profiling in blood samples | Up to 24 months
  Whole-genome methylation analysis and locus specific analysis of selected stress related genes, will be conducted to investigate early, intermediate and long-term epigenetic changes due to the intervention.
Telomere profiling in blood samples | Up to 24 months
  Whole-genome methylation analysis and locus specific analysis of selected stress related genes, will be conducted to investigate telomere length
Microbiota | 0-6 hours, 72 hours, 3-4 months, 12 and 24 months. Mother is tested at 0-6 hours and partner with skin swabs at 0-6 hours.
  The child's colonization with bacteria is identified by DNA-analysis from stool samples, nasal and skin swabs, compared with parents (mother is tested by vaginal, rectal, nasal and skin swabs.
Maturation of EEG-pattern | Postnatal day 4-10 and postmenstrual age of 40-42 weeks
Structural and functional maturation of the infant brain | At term age
  Magnetic Resonance Imaging scans will be performed with a 3 Tesla machine. Three-dimensional and diffusion sequences as well as functional MRI (fMRI) sequences will be performed in order to examine structural and functional maturation respectively. Structural sequences are used to study the different tissues of the brain; diffusion images give information about the connections of the brain (white matter) and fMRI gives information on how the brain integrates information to perform a specific function.
Maternal brain responsiveness | At 4 months
  The maternal brain responses will be evaluated by using structural and functional magnetic resonance imaging to measure structural changes on social, emotional and behavioural networks as well as the cerebral response of mothers viewing neutral, happy and distress face images of their own infant, along with a matched unknown infant. We will use a 3 Tesla machine. We will study cortical and subcortical networks related with the emotional, social and behavioral responses involving the mother-child interactions and responses, such as the insula, the cingulate cortex, the precentral gyrus, the right orbital gyrus, the inferior, middle and superior frontal gyrus the fusiform gyrus, supramarginal gyrus, the superior parietal gyrus, the inferior temporal gyrus, and basal ganglia among others.
Bonding and interaction between parent and child | At 3-4 months and at 12 and 24 months.
  A videotaped mother-infant interaction session will be assessed through with the Parent-Child Early Relational Assessment (PCERA)
Bonding and interaction between parent and child | At 3-4 months
  A videotaped mother-infant interaction session will be assessed through the "Still Face situation"
Parents' experiences | Up to 12 months
  Parents will fill in the following questionnaire: State-Trait Anxiety Index(STAI)
Parents' experiences | Up to 12 months
  Parents will fill in the following questionnaire: Swedish Parenting Questionnaire (SPSQ)
Parents' experiences | Up to 12 months
  Parents will fill in the following questionnaire: Edinburgh postnatal Depression Scale (EPDS)
Maternal-Child physiological attunement in stress regulation | In the morning and in the evening at the day of discharge, At the day of discharge before and after diaper change, at 3-4 months, at the same day as Still Face-test before and after, at 12 months.
  Saliva Cortisol both mother and child
Neuro Behaviour of Child | At term age, at 3-4, 12 and 24 months
  According to records and to questionnaires for example Infant Behavior Questionnaire (IBQ)
Neuro Behaviour of Child | At term age, at 3-4, 12 and 24 months
  According to records and to questionnaires for example Bayley Scales
Neuro Behaviour of Child | At term age, at 3-4, 12 and 24 months
  According to records and to questionnaires for example Ages and Stages Questionnaire (ASQ)

CONTACTS AND LOCATIONS:
Overall Officials: Björn Westrup, MD,PhD, Study Chair — Department of Women´s and Children´s Health, Karolinska Institutet, Stockholm, Sweden; Siren Rettedal, MD, PhD, Principal Investigator — Stavanger University Hospital, Stavanger, Norway; Wibke Jonas, Ass prof, Principal Investigator — Department of Women´s and Children´s Health, Karolinska Institutet, Stockholm, Sweden
Locations (2):
- Stavanger University Hospital, Stavanger, Norway
- Department of Women´s and Children´s Health, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lillieskold S, Lode-Kolz K, Rettedal S, Lindstedt J, Linner A, Markhus Pike H, Ahlqvist-Bjorkroth S, Aden U, Jonas W. Skin-to-Skin Contact at Birth for Very Preterm Infants and Mother-Infant Interaction Quality at 4 Months: A Secondary Analysis of the IPISTOSS Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2344469. doi: 10.1001/jamanetworkopen.2023.44469. PMID 38032643
- [Derived] Linner A, Westrup B, Lode-Kolz K, Klemming S, Lillieskold S, Markhus Pike H, Morgan B, Bergman NJ, Rettedal S, Jonas W. Immediate parent-infant skin-to-skin study (IPISTOSS): study protocol of a randomised controlled trial on very preterm infants cared for in skin-to-skin contact immediately after birth and potential physiological, epigenetic, psychological and neurodevelopmental consequences. BMJ Open. 2020 Jul 6;10(7):e038938. doi: 10.1136/bmjopen-2020-038938. PMID 32636292